CLINICAL TRIAL: NCT04897100
Title: Outcome and Complications After Percutaneous Needle Versus Blade Achilles Tenotomy in Clubfoot Treated With the Ponseti Method
Brief Title: Outcome After Needle vs Blade Achilles Tenotomy in Clubfoot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indus Hospital and Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRD_IRB_2020_03_011
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Club Foot; Achilles Tendon Surgery
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needle tenotomy (Experimental): Patient will receive an Achilles tendon tenotomy using a 22G needle when randomized into the needle group. Follow-up to measure dorsiflexion and register complications will be assured at 3 weeks and 3 months.
  Interventions: Procedure: Achilles tendon tenotomy
- Blade tenotomy (Active Comparator): Patient will receive an Achilles tendon tenotomy using a 11 blade when randomized into the needle group. Follow-up to measure dorsiflexion and register complications will be assured at 3 weeks and 3 months.
  Interventions: Procedure: Achilles tendon tenotomy

INTERVENTIONS:
Procedure: Achilles tendon tenotomy — Achilles tendon tenotomy during Ponseti treatment for clubfoot

SUMMARY:
Achilles tendon tenotomy is an integral part of the Ponseti method, aimed at correcting residual equinus after correction of the adductus deformity. Tenotomy rates ranging from 63-95% after full cycle of castings have been reported in literature. Percutaneous tenotomy is the gold standard, which can usually be performed in an out-patient setting under local anesthesia using a scalpel blade. A complication rate of 2% (mainly neurovascular injury)has been reported in literature, with accidental sectioning of the peroneal artery being the most common. Development of a pseudo-aneurysm after accidental sectioning of the peroneal artery has been reported in a case report; this delayed further clubfoot treatment.

Percutaneous needle tenotomy has been described by some authors as an alternative technique with very favorable results in a population before walking age. This technique use a large-gauge (16-19 G) needle to percutaneously cut the Achilles tendon. Although bleeding has been reported following this technique with similar rates as for the percutaneous blade technique, no major complications have been reported as yet using the needle technique.

We would like to compare the clinical outcomes and complication rates of both techniques, supporting our hypothesis that both techniques are equally safe and have the same success rate.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic clubfoot.
* Age less than or equal to 36 months at the time of tenotomy.
* Enrolled at the Pehla Qadam clinic at The Indus Hospital in Karachi.
* Fully corrected Adductus deformity with residual equinus after a full casting cycle.
* Completing routine follow up for 3 months post tenotomy.

Exclusion Criteria:

* Refusal of parents to enroll child into this study.
* Syndromic clubfoot.
* Previous treatment for clubfoot (surgical or non-surgical) received.
* Underlying medical conditions unrelated to clubfoot that may serve as a contra-indication, this decision will be left on the discretion of the treating orthopedic surgeon

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 244 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2023-09-02 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
Dorsiflexion | 3 months
  Ankle dorsiflexion measured in degrees

SECONDARY OUTCOMES:
Complications | 3 months
  Post-op complications due to tenotomy

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor Khan, Principal Investigator — Indus Hospital and Health Network
Locations (1):
- Indus Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The participant data will be made available in an anonymous manner as a supplement to the final publication
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Pigeolet M, Ghufran Syed J, Ahmed S, Chinoy MA, Khan MA. A single-center, single-blinded, randomized, parallel-group, non-inferiority trial to compare the efficacy of a 22-gauge needle versus a 15 blade to perform an Achilles tendon tenotomy in 244 clubfeet-study protocol. Trials. 2023 Oct 31;24(1):701. doi: 10.1186/s13063-023-07728-9. PMID 37907927